CLINICAL TRIAL: NCT01111682
Title: Hypertonic Saline vs. Mannitol for Elevated Intercranial Pressure
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: A significant reduction in head injuries coupled with more frequent use of crainectomy reduced the number of potential subjects.
Sponsor: University of Cincinnati (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Shutter-2010-01
Record Dates: First submitted 2010-04-22; First posted 2010-04-27 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Traumatic Brain Injury; Elevated Intracranial Pressure
Keywords: traumatic brain injury; hypertonic saline therapy; intracranial pressure
MeSH Terms: conditions — Brain Injuries, Traumatic; Intracranial Hypertension | interventions — Mannitol; Saline Solution, Hypertonic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mannitol (Active Comparator): 0.9% normal saline infusion and boluses of mannitol
  Interventions: Drug: Mannitol
- Hypertonic Saline (Active Comparator): 3% hypertonic saline continuous infusion, with intermittent boluses as needed
  Interventions: Drug: Hypertonic Saline

INTERVENTIONS:
Drug: Mannitol — 0.9% normal saline infusion and boluses of mannitol
  Arms: Mannitol
Drug: Hypertonic Saline — 3% hypertonic saline continuous infusion, with intermittent boluses as needed
  Arms: Hypertonic Saline

SUMMARY:
This study examines the role of osmotic agents in controlling brain swelling in brain injured individuals. Two osmotic agents -- mannitol and hypertonic saline -- are in common use, and they will be compared in the context of a randomized clinical trial. The goal is to determine if these agent differ in their ability to control episodes of brain swelling.

DETAILED DESCRIPTION:
This single-center, randomized, open label trial will compare (i) 0.9% normal saline infusion and boluses of mannitol (control group) with (ii) 3% hypertonic saline, with intermittent boluses as needed, to treat elevated intracranial pressure (ICP) following severe traumatic brain injury.

Patients will be randomized to one of the two study arms following placement of an ICP monitor. Raised ICP will be defined as an ICP greater than 20 mmHG for 20 minutes or longer. In the event of such an event, the appropriate treatment will be administered.

The primary endpoint will be success in ICP control, operationalized as the proportion of time during which ICP is less than or equal to 20 mmHg during the first 120 hours following initiation of monitoring. Secondary endpoints include therapy intensity level, incidence of pre-determined severe adverse events, and long-term outcomes measured at 3 and 6 months post-injury.

ELIGIBILITY:
Inclusion Criteria:

* closed traumatic brain injury
* either (i) GCS score 3-8 (inclusive), or (ii) GCS motor score of 5 or less AND abnormal admission CT scan showing intracranial pathology
* hemodynamically stable with systolic blood pressure greater than 90 mmHg
* at least 1 reactive pupil
* age between 18y and 70y (inclusive)
* INR less than 1.5

Exclusion Criteria:

* actively on hypertonic saline or mannitol
* hypernatremia (>145 meq/L)
* anuric or with creatinine greater than or equal to 2.5
* known seizure disorder
* penetrating head trauma
* suspected anoxic events
* history of, or CT confirmation of, previous brain injury
* any injury that, in the opinion of the Principal Investigator, has a high likelihood of death with the first 72 hours post-injury
* any treatment, condition, or injury that contraindicates treatment with hypertonic saline

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-04; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Proportion of time during which ICP is less than or equal to 20 mmHg during the first 120 hours following initiation of ICP monitoring. In the case where a patient is weaned from infusion, full ICP control will be assumed. | 120 hours post initiation of monitoring
  ICP will be recorded continuously and the proportion of time during which ICP is uncontrolled will be calculated. Specifically, this will be measured as any period during which ICP > 20 mmHg for 600 seconds or longer.

SECONDARY OUTCOMES:
Therapy Intensity Level (TIL), reflecting the amount and duration of therapy required to control ICP. TIL incorporates, among others, variables such as degree of head elevation, level of sedation, volume of CSF drainage, and hypocapnia. | Daily
Long-term outcomes measured by Disability Rating Scale and Glasgow Outcome Scale-Extended | 3 and 6 months post-injury
Incidence of pre-determined severe adverse events (SAEs): brain hypoxia, delayed decompression, pulmonary edema, renal failure, respiratory complications, seizures, systemic hypoxia, and uncontrollable ICP | Each occurence of an SAE during the patient's hospital stay will be recorded.
  For each patient, we will count the number of SAEs in each category. Total SAEs by category and average number of SAEs per patient will be compared between the two study treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Lori Shutter, MD, Principal Investigator — Department of Neurology College of Medicine University of Cincinnati
Locations (1):
- University Hospital, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Zornow MH. Hypertonic saline as a safe and efficacious treatment of intracranial hypertension. J Neurosurg Anesthesiol. 1996 Apr;8(2):175-7. doi: 10.1097/00008506-199604000-00021. No abstract available. PMID 8829566
- [Background] Doyle JA, Davis DP, Hoyt DB. The use of hypertonic saline in the treatment of traumatic brain injury. J Trauma. 2001 Feb;50(2):367-83. doi: 10.1097/00005373-200102000-00030. No abstract available. PMID 11242309
- [Background] Qureshi AI, Suarez JI. Use of hypertonic saline solutions in treatment of cerebral edema and intracranial hypertension. Crit Care Med. 2000 Sep;28(9):3301-13. doi: 10.1097/00003246-200009000-00032. PMID 11008996
- [Background] Gunnar W, Jonasson O, Merlotti G, Stone J, Barrett J. Head injury and hemorrhagic shock: studies of the blood brain barrier and intracranial pressure after resuscitation with normal saline solution, 3% saline solution, and dextran-40. Surgery. 1988 Apr;103(4):398-407. PMID 2451302
- [Background] Ogden AT, Mayer SA, Connolly ES Jr. Hyperosmolar agents in neurosurgical practice: the evolving role of hypertonic saline. Neurosurgery. 2005 Aug;57(2):207-15; discussion 207-15. doi: 10.1227/01.neu.0000166533.79031.d8. PMID 16094147